CLINICAL TRIAL: NCT06575764
Title: The Heart Priority Programme for Patients at Risk of Dropout From Cardiac Rehabilitation - a Development- and Feasibility Study
Brief Title: The Heart Priority Programme for Cardiac Patients at Risk of Dropout From Cardiac Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defactum, Central Denmark Region (Other Government)
Collaborators: University of Aarhus (Other); Aarhus Municipality, Denmark (Other); Viborg Municipality, Denmark (Unknown); Ringkøbing-Skjern municipality, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: The Heart Priority Programme
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiac Rehabilitation; Complex intervention; Co-production; Intervention development; Feasibility study; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart priority Programme (Experimental): The Heart Priority Programme was developed to supplement standardised cardiac rehabilitation to reduce dropouts among cardiac patients at risk of dropout due to being in a vulnerable situation
  Interventions: Other: The Heart Priority Programme

INTERVENTIONS:
Other: The Heart Priority Programme — The programme is delivered by the Cardiac Rehabilitation (CR) team. It consist of two main parts: 1) an evidence-based identification form to identify patients at risk of dropout due to being in a vulnerable situation and 2) an add-on intervention to standard CR targeted these patients. The add-on intervention encompasses three core elements: 1) Assigning a contact person with specific responsibilities, 2) Systematically communicating patient information to colleagues in the CR team and 3) Systematic follow-up

SUMMARY:
The goal of this study is to develop The Heart Priority programme, a supplement to standardised cardiac rehabilitation (CR) aimed at identifying and supporting cardiac patients at risk of dropout due to being in a vulnerable situation. Additionally, the study aims to test the programme through a feasibility study.

The programme comprises two main parts: 1) an evidence-based identification form to identify patients at risk of dropout from CR due to being in a vulnerable situation and 2) an add-on intervention targeted these patients.

The study will be guided by the Medical Research Council's framework for developing and evaluating complex interventions (MRC). The development follows an iterative three-stage process guided by the framework for co-producing and prototyping of healthcare interventions. Stage 1 is preparation by considering the knowledgebase. Building on this knowledge, stage 2 and 3 includes a co-production and prototyping process, aiming to develop, field test and adapt the programme, deemed ready for feasibility testing.

The feasibility study will be designed as a single-arm follow-up study conducted in two community health care centres in Denmark. Process data will be collected continuously over a six-months period and at the study's conclusion, focussing on three dimensions: implementation (reach and fidelity), acceptability, and mechanism of impact.

DETAILED DESCRIPTION:
Despite advancements in reducing cardiovascular disease, heart disease remains a significant health issue. Cardiac rehabilitation (CR) is crucial for recovery, with evidence showing its positive impact on morbidity, mortality, and functioning. However, dropout rates, especially among patients in a vulnerable situation, are high due to social inequalities and lack of tailored interventions. To implement interventions for individuals in a vulnerable situation, it is necessary to: 1) identify the target group and 2) develop an intervention tailored to the group. There is currently no such intervention within the field of CR. Therefore, we developed, and feasibility tested the Heart Priority Programme aiming to reduce dropouts in cardiac rehabilitation among patients in a vulnerable situation.

The purpose is to develop the Heart Priority Programme in close collaboration with stakeholders and subsequently conduct a feasibility study in community healthcare services within the Central Denmark Region.

The study follows the Medical Research Council's framework for developing complex interventions, focusing on the development and feasibility phases.

First a development study will be conducted. The development of the Heart Priority Programme will follow a three-stage iterative process, including evidence review, stakeholder consultations, co-production of intervention content, and prototyping involving close collaboration between cardiac patients, healthcare professionals, and researchers. The Heart Priority Programme encompasses two main parts: 1) an evidence-based identification form to identify patients being in a vulnerable situation (professional tool to be used during the initial consultation) and 2) an add-on intervention to supplement standard CR targeted these patients.

Subsequently, a feasibility study designed as a single-arm follow-up study will be conducted in two community healthcare services in Central Denmark Region. The programme is delivered by the CR team. The evidence-based identification form will be used for all cardiac patients referred to CR and fulfilled during the initial consultation. If the healthcare professional identifies a patient at risk of dropout due to being in a vulnerable situation this patient will receive the add-on intervention targeted these patients. The add-on intervention encompasses three core elements:

1. Assigning a contact person with specific responsibilities (e.g., ensure the patient feels safe and welcome at the first session, and acting as a contact in case of cancellation)
2. Systematically communicating patient information to colleagues in the CR team
3. Systematic follow-up (e.g., maintaining continuous contact in case of cancellation/absence, and ongoing follow-up).

The add-intervention will be described in detailed in accordance with the Template for Intervention Description and Replication (TIDieR)

Both quantitative (data from the identification form) and qualitative methods (data from feedback meetings with healthcare professionals) will be used to collect data. Process data will be collected continuously over a six-months period and at the study's conclusion, focussing on three dimensions: implementation (reach and fidelity), acceptability, and mechanism of impact. Descriptive statistics will be used to analyse implementation data, while content-driven analysis will be applied to assess acceptability and mechanisms of impact. Based on clinical and research judgment, a convenience sample of at least 150 cardiac patients referred to CR was deemed sufficient to adequately represent the target population and provide data for the feasibility study.

According to Danish legislation and the Act on Biomedical Research Ethics Committee System in Denmark, research without human biological material does not require approval from an ethics committee (§14 Section 2). The study was registered and approved by the Data Protection Agency of Central Denmark Region (1-16-02-121-24). Cardiac patients and healthcare professionals provide written informed consent to participate in the co-production process, like participants in the feasibility test.

If the feasibility study yields promising results, a larger-scale study will be conducted to evaluate the Heart Priority Programme's overall impact on dropout rates in cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute coronary syndrome
* age >18 years
* patients referred to CR in community healthcare services
* patients living in Central Denmark Region
* patients at risk of dropout due to being in a vulnerable situation.

Exclusion Criteria:

* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Implementation (reach and fidelity) | Six months
  Evaluate: 1)The extent to which the target group encounters the programme (reach) and 2) Whether the programme was delivered as intended (fidelity)

SECONDARY OUTCOMES:
Acceptability | Six months
  Evaluate the CR teams' view on the programme
Mechanisms of impact | Six months
  Evaluate how the CR teams respond to and interact with the programme

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ibsen, PhD, Principal Investigator — Defactum, Central Denmark Region; Thomas Maribo, PhD, Study Chair — Defactum, Central Denmark Region and Aarhus University
Locations (3):
- Denmark (3):
  - Aarhus Municipality, Aarhus
  - Ringkøbing-Skjern Municipality, Ringkøbing
  - Viborg Municipality, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur J Prev Cardiol. 2022 Feb 19;29(1):5-115. doi: 10.1093/eurjpc/zwab154. No abstract available. PMID 34558602
- [Background] Cowie A, Buckley J, Doherty P, Furze G, Hayward J, Hinton S, Jones J, Speck L, Dalal H, Mills J; British Association for Cardiovascular Prevention and Rehabilitation (BACPR). Standards and core components for cardiovascular disease prevention and rehabilitation. Heart. 2019 Apr;105(7):510-515. doi: 10.1136/heartjnl-2018-314206. Epub 2019 Jan 30. PMID 30700518
- [Background] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536
- [Background] Santiago de Araujo Pio C, Chaves GS, Davies P, Taylor RS, Grace SL. Interventions to promote patient utilisation of cardiac rehabilitation. Cochrane Database Syst Rev. 2019 Feb 1;2(2):CD007131. doi: 10.1002/14651858.CD007131.pub4. PMID 30706942
- [Background] Turk-Adawi KI, Grace SL. Narrative review comparing the benefits of and participation in cardiac rehabilitation in high-, middle- and low-income countries. Heart Lung Circ. 2015 May;24(5):510-20. doi: 10.1016/j.hlc.2014.11.013. Epub 2014 Nov 29. PMID 25534902
- [Background] Resurreccion DM, Motrico E, Rigabert A, Rubio-Valera M, Conejo-Ceron S, Pastor L, Moreno-Peral P. Barriers for Nonparticipation and Dropout of Women in Cardiac Rehabilitation Programs: A Systematic Review. J Womens Health (Larchmt). 2017 Aug;26(8):849-859. doi: 10.1089/jwh.2016.6249. Epub 2017 Apr 7. PMID 28388314
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Hawkins J, Madden K, Fletcher A, Midgley L, Grant A, Cox G, Moore L, Campbell R, Murphy S, Bonell C, White J. Development of a framework for the co-production and prototyping of public health interventions. BMC Public Health. 2017 Sep 4;17(1):689. doi: 10.1186/s12889-017-4695-8. PMID 28870192
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] O'Cathain A, Hoddinott P, Lewin S, Thomas KJ, Young B, Adamson J, Jansen YJ, Mills N, Moore G, Donovan JL. Maximising the impact of qualitative research in feasibility studies for randomised controlled trials: guidance for researchers. Pilot Feasibility Stud. 2015 Sep 7;1:32. doi: 10.1186/s40814-015-0026-y. eCollection 2015. PMID 27965810
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Derived] Ibsen C, Katholm KK, Jakobsen A, Eriksen GB, Lysdal L, Nielsen UK, Ravn MB, Maribo T. Reducing dropout rates in cardiac rehabilitation among cardiac patients in a vulnerable situation: systematic development and feasibility testing of the Heart Priority Programme. BMC Health Serv Res. 2024 Dec 18;24(1):1579. doi: 10.1186/s12913-024-12073-x. PMID 39695726
- See also: Danish Health Authority. National Clinical Guideline On Cardiac Rehabilitation, 2015 — https://www.sst.dk/da/udgivelser/2015/~/media/401919781C684EE9AAE544EB5E76847B.ashx